CLINICAL TRIAL: NCT01531998
Title: An Open Label, Single-Arm, Phase 1b/2 Study of the Safety and Efficacy of Combination Treatment With Lenalidomide, Bortezomib, Dexamethasone and Siltuximab (CNTO 328) in Subjects With Newly Diagnosed, Previously Untreated Multiple Myeloma Requiring Systemic Chemotherapy
Brief Title: Lenalidomide/Bortezomib/Dexamethasone & CNTO 328 in Transplant Eligible Newly Diagnosed Multiple Myeloma (MM)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Janssen Services, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-0073; NCI-2012-00218 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-02-09; First posted 2012-02-13 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Myeloma
Keywords: Myeloma; Multiple Myeloma; MM; Newly diagnosed; Lenalidomide; CC-5013; Revlimid; Bortezomib; Velcade; LDP-341; MLN341; PS-341; Siltuximab; CNTO 328; Anti-IL-6 Antibody; Dexamethasone; Decadron; M. D. Anderson Symptom Inventory Module; MDASI-MM; Questionnaires; Surveys
MeSH Terms: conditions — Neoplasms, Plasma Cell; Multiple Myeloma | interventions — Lenalidomide; Bortezomib; siltuximab; Dexamethasone; Calcium Dobesilate; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Siltuximab + Bortezomib + Lenalidomide (Experimental): Induction: Lenalidomide 25 mg orally Days 1-14; Bortezomib 1.3 mg/m2 intravenous Days 1, 4, 8 and 11; Dexamethasone 20 mg orally Days 1, 2, 4, 5, 8, 9, 11, 12. Siltuximab 11 mg/kg intravenous Day 1.
  If delayed transplant, induction therapy continued up to 2 cycles beyond achieving a CR/nCR (minimum of 4 cycles of therapy and a maximum of 8 cycles of therapy) and then transition to maintenance regimen described below.
  Maintenance therapy: Lenalidomide at last tolerated dose Day 1-21 every 28 days for up to 12 months and then may be reduced to 10 mg.
  Siltuximab 11 mg/kg intravenous every 21 days, or maximum tolerated dose from induction therapy. Bortezomib at last tolerated dose Day 1 and Day 8 Dexamethasone at last tolerated dose or 20 mg weekly.
  Interventions: Drug: Lenalidomide; Drug: Bortezomib; Drug: Siltuximab; Drug: Dexamethasone; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Lenalidomide — Induction Phase: 25 mg by mouth daily on Days 1-14. Maintenance Phase: at last tolerated dose from Induction Phase day 1-21 every 28 days for up to 12 months and then may be reduced to 10 mg.
  Other Names: CC-5013; Revlimid
Drug: Bortezomib — Induction Phase: 1.3 mg/m2 by vein daily on Days 1, 4, 8 and 11.
  Maintenance Phase: 1.3 mg/m2 by vein or last tolerated dose on Day 1 and Day 8.
  Other Names: Velcade; LDP-341; MLN341; PS-341
Drug: Siltuximab — Induction Phase Starting Dose: 11 mg/kg by vein on Day 1.
  Maintenance Phase: 11 mg/kg intravenous every 21 days, or maximum tolerated dose from induction therapy.
  Other Names: CNTO 328; Anti-IL-6 Antibody
Drug: Dexamethasone — Induction Phase: 20 mg by mouth on Days 1, 2, 4, 5, 8, 9, 11, 12.
  Maintenance Phase: 20 mg by mouth on Days 1, 2, 4, 5, 8, 9, 11, 12. If participant still on Dexamethasone, when entering Maintenance Phase, dose reduced to 20 mg a week.
  Other Names: Decadron
Behavioral: Questionnaires — M. D. Anderson Symptom Inventory Module (MDASI-MM) completed Day 1, Day 8 of Cycle 1 - 8, and on Day 1 of Cycle 9 and beyond.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of Siltuximab that can be given in combination with Velcade (bortezomib), Revlimid (lenalidomide), and dexamethasone to patients with MM. The safety of this drug combination will also be studied.

DETAILED DESCRIPTION:
The Study Drugs:

Siltuximab is designed to block IL-6, which is a protein that plays an important role in the survival of myeloma cancer cells. This may slow the growth of cancer cells or cause the cancer cells to die.

Bortezomib is designed to block a protein that plays a role in cell function and growth. This may cause cancer cells to die.

Lenalidomide is designed to kill the myeloma cells and may change the body's immune system. It may also interfere with the development of tiny blood vessels that help support tumor growth. This may slow the growth of cancer cells.

Dexamethasone is a corticosteroid that is similar to a natural hormone made by your body. Dexamethasone is often given to MM patients in combination with other chemotherapy to treat cancer.

Study Groups:

If you are found to be eligible to take part in this study, based on when you join the study you will be enrolled in the Phase I or Phase II portion. If you are in Phase I, you will be assigned to a dose level of Siltuximab based on when you join this study. Up to 2 dose levels of Siltuximab will be tested. Three (3) to 6 participants will be enrolled at each dose level. The first group of participants will receive the highest dose level. If intolerable side effects are seen in the first group, the next group will receive a lower dose.

All participants will receive the same dose level of bortezomib, lenalidomide, and dexamethasone.

After the highest tolerable dose level is found, up to an extra 54 participants will receive the study drugs at this dose level in the Phase II part of the study.

Study Drug Administration:

Induction Therapy - Each cycle is 21 days. On Days 1, 4, 8, and 11 of Cycle 1 up to Cycle 8 (induction therapy), you will receive bortezomib through a needle under the skin or by vein over 3-5 seconds.

On Days 1-14 of every cycle, you will take lenalidomide by mouth 1 time each day. Swallow lenalidomide capsules whole with 1 cup (about 8 ounces) of water. Do not break, chew, or open the capsules.

On Day 1 of every cycle, you will receive Siltuximab by vein over 1 hour.

On Days 1, 2, 4, 5, 8, 9, 11, and 12 of Cycles 1-8 (induction therapy), you will take dexamethasone by mouth 1 time a day. After 8 cycles, you may continue to take dexamethasone if the doctor thinks it is needed. Dexamethasone should be taken with food.

You can take the study drugs any time during the day but you should take them at the same time every day.

If you miss a dose of lenalidomide, take it as soon as you remember on the same day. If you miss taking your dose for the entire day, take your regular dose the next scheduled day (do NOT take double your regular dose to make up for the missed dose). If you take more than the prescribed dose of lenalidomide, you should seek emergency medical care if needed and contact the study staff right away.

You will be given a study drug dosing calendar for each cycle to record the lenalidomide and dexamethasone you will be taking at home. Please bring the dosing calendar and pill bottles to your study visit at the beginning of each new cycle.

If the doctor thinks it is in your best interest, you may have a stem cell transplant anytime after 4 cycles of induction therapy You will sign a separate consent form that will describe the procedure and the risks in detail.

Maintenance Phase - Each cycle is 28 days. If you want to delay the stem cell transplant, after 4-8 cycles, you will begin the maintenance phase.

During the maintenance phase:

* You will take lenalidomide on Days 1-21 of each cycle.
* You will take dexamethasone by mouth once a week.
* You will receive Siltuximab by vein on Day 1 of every cycle.

Study Visits:

On Day 1 of Cycle 1:

* You will have a physical exam, including measurement of your height, weight and vital signs.
* Your medical history will be updated.
* You will be asked to list any drugs you may be taking and if you have had any side effects.
* Your performance status will be recorded.
* You will have an ECG.
* You will complete 2 questionnaires about your day-to-day activities and quality of life. They should take about 5 minutes each to complete.
* If you are able to become pregnant, you will have a blood or urine (about 1 teaspoon) pregnancy test.
* Blood (about 2 tablespoons) will be drawn to measure protein levels, which may help researchers learn more about how to better treat myeloma.

On Day 1 of Cycles 2-8:

* You will have a physical exam, including measurement of your height, weight and vital signs.
* Your performance status will be recorded.
* You will be asked to list any drugs you may be taking and if you have had any side effects.
* Blood (about 5 tablespoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) and/or urine will be collected to check the status of the disease. If urine is collected, you will collect the urine over 24 hours. You will be provided with a container to collect the urine in.
* Blood (about 2 tablespoons) will be drawn to measure protein levels, which may help researchers learn more about how to better treat myeloma.
* You will complete the questionnaire about your day-to-day activities
* If you are able to become pregnant, you will have a blood or urine (about 1 teaspoon) pregnancy test.

On Days 4 of Cycles 1-8:

-Blood (about 4 tablespoons) will be drawn for routine tests.

On Day 8 of Cycle 1:

-You will have a bone marrow aspirate to better understand how the drugs are affecting the myeloma. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

On Days 8 of Cycles 1-8:

-Blood (about 4 tablespoons) will be drawn for routine tests. During Cycle 1, this routine blood draw will include a pregnancy test if you are able to become pregnant.

On Day 11 of Cycles 1-8:

-Blood (about 4 tablespoons) will be drawn for routine tests.

At the end of induction therapy (or if you are going to have a stem cell transplant, at the end of Cycle 4):

* You will have a physical exam.
* You will be asked to list any drugs you may be taking and if you have had any side effects.
* Blood (about 5 tablespoons) and urine will be collected for routine tests.
* You will have a skeletal survey to check the status of the disease.
* If the disease completely responds to the study drugs, you will have a bone marrow aspiration and/or biopsy to check the status of the response.

On Day 1 of Cycles 9 and beyond (Maintenance Therapy):

* You will have a physical exam, including measurement of your vital signs, height, and weight.
* Your performance status will be recorded.
* You will be asked to list any drugs you may be taking and if you have had any side effects.
* Blood (about 4 tablespoons) will be drawn for routine tests.
* Blood (about 1 teaspoon) and/or urine will be collected to check the status of the disease. If urine is collected, you will collect the urine for 24 hours. You will be provided with a container to collect the urine in.
* If the doctor thinks it is needed, you will have a skeletal survey to check the status of the disease.
* If the doctor thinks it is needed, you will have an MRI scan or CT scan to check the status of the disease.
* Blood (about 2 tablespoons) will be drawn to measure protein levels, which may help researchers learn more about how to better treat myeloma.
* You will complete the questionnaires about your day-to-day activities and quality of life.

Pregnancy Tests:

During induction therapy, if you are a woman who is able to become pregnant and you have regular or no periods, you will have a blood (about 1 tablespoon) or urine pregnancy test weekly for the first 21 days and then every 21 days while on therapy (including breaks in therapy). If you are a woman who is able to become pregnant and your cycles are irregular, you will have a blood (about 1 tablespoon) or urine pregnancy test weekly for the first 21 days during then every 11-14 days while on therapy (including breaks in therapy).

During maintenance therapy, if you are a woman who is able to become pregnant and have regular or no menstruation, you must have a pregnancy test every 28 days while on therapy (including breaks in therapy). If you are a woman who is able to become pregnant and your cycles are irregular, you will have a blood (about 1 tablespoon) or urine pregnancy test every 14 days (+/-1 day) and every 28 days.

Length of Study:

You may stay on study for as long as the disease does not get worse, you have not experienced intolerable side effects, and if the study doctor thinks it is in your best interest.

End-of-Treatment Visit:

Within 1 month after the last dose of study drugs, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* Your performance status will be recorded.
* You will be asked to list any drugs you may be taking and if you have had any side effects.
* You will have a physical exam, including measurement of your height and weight.
* You will have a skeletal survey.
* You will have a bone marrow biopsy to check the status of the disease.
* Blood (about 4 tablespoon) and urine will be collected for routine tests.

Long-Term Follow-Up:

If you go off study for reasons other then the disease getting worse, blood (about 5 tablespoons) will be drawn for routine tests. This will done every 3 months for the first 2 years, every 6 months for Years 3 and 4, and yearly for Years 5 and 6. The long term visits will be to check disease status, survival, long term side effects, and secondary cancers.

This is an investigational study. Siltuximab is not FDA approved or commercially available. It is only being used for research at this time. Bortezomib is FDA approved and commercially available for the front-line treatment of MM. Lenalidomide is FDA approved and commercially available for the treatment of certain types of myelodysplastic syndrome and for use with dexamethasone for patients with MM who have received at least 1 therapy. The use of this drug combination to treat MM is investigational.

Up to 11 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 1. Multiple Myeloma Diagnosis: Subject was previously diagnosed with multiple myeloma by the International Myeloma Foundation 2003 Diagnostic Criteria: IMF Diagnostic Criteria: DIAGNOSTIC CRITERIA: ALL 3 REQUIRED 1. Monoclonal plasma cells in the bone marrow > 10% and/or presence of a biopsy-proven plasmacytoma 2. Monoclonal protein present in the serum and/or urine * 3. Myeloma-related organ dysfunction (1 or more) ** ; [C] Calcium elevation in the blood S. Calcium >10.5 mg/l or upper limit of normal ; [R] Renal insufficiency ; [A] Anemia Hemoglobin < 10 g/dl or 2 g < normal ; [B] Lytic bone lesions or osteoporosis ***
2. Continuation from Inclusion # 1: *If no monoclonal protein is detected (non-secretory disease), then > 30% monoclonal bone marrow plasma cells and/or a biopsy-proven plasmacytoma required ** A variety of other types of end organ dysfunctions can occasionally occur and lead to a need for therapy. Such dysfunction is sufficient to support classification of myeloma if proven to be myeloma related. *** If a solitary (biopsy-proven) plasmacytoma or osteoporosis alone (without fractures) are the sole defining criteria, then > 30% plasma cells are required in the bone marrow.
3. Patient must not have been previously treated with any prior systemic therapy for the treatment of multiple myeloma. Prior treatment of hypercalcemia or spinal cord compression with corticosteroids does not disqualify the patient (the dose should not exceed the equivalent of 160 mg of dexamethasone in a 2 week period). Bisphosphonates are permitted
4. Patients treated with local radiotherapy with or without concomitant exposure to steroids, for pain control or management of cord/nerve root compression, are eligible. One week must have lapsed since last date of radiotherapy, which is recommended to be a limited field. Patients who require concurrent radiotherapy should have start of the protocol therapy (Cycle 1 Day 1) deferred until the radiotherapy is completed and one week have passed since the last date of therapy.
5. Voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to future medical care.
6. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test with a sensitivity of at least 50 milli-International unit (mIU)/mL 10 - 14 days prior to therapy and repeated again within 24 hours of prescribing lenalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy. All patients must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure.
7. Age >/= 18 years at the time of signing Informed Consent.
8. All necessary baseline studies for determining eligibility must be obtained within 28 days prior to enrollment.
9. Subject has a Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
10. All study participants must be registered into the mandatory RevAssist program, and be willing and able to comply with the requirements of RevAssist.
11. Able to take aspirin (81 or 325 mg) daily as prophylactic anticoagulation (patients intolerant to ASA may use warfarin or low molecular weight heparin).
12. Subject must be able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Patient has >/=Grade 2 peripheral neuropathy on clinical examination within 14 days before enrollment.
2. Renal insufficiency (Creatinine Clearance <30 mL/min by Cockcroft -Gault formula).
3. Subjects with evidence of mucosal or internal bleeding and/or platelet refractory (i.e., unable to maintain a platelet count >/= 50,000 cells/mm^3).
4. Subjects with an absolute neutrophil count (ANC) < 1000 cells/mm^3. Growth factors may not be used to meet ANC eligibility criteria.
5. Total bilirubin > 1.5 mg/dL
6. Subjects with a hemoglobin < 8.0 g/dL (Transfusion are permitted).
7. AST (SGOT and ALT (SGPT) >/= 2 x upper limit of normal (ULN)
8. Myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
9. Clinically relevant active infection requiring intravenous antibiotics
10. Serious co-morbid medical conditions such as uncontrolled chronic obstructive or chronic restrictive pulmonary disease, and cirrhosis.
11. Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the subject at unacceptable risk if he/she were to participate in the study.
12. Female subject is pregnant or breast-feeding.
13. Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
14. Uncontrolled diabetes mellitus (Fasting Blood Sugar > 400 mg/dl despite medical treatment)
15. Hypersensitivity to acyclovir or similar anti-viral drug
16. Known history of POEMS syndrome (plasma cell dyscrasia with polyneuropathy, organomegaly, endocrinopathy, monoclonal protein (M-protein) and skin changes).
17. Patients with known history of HIV, Hep B and C.
18. Hypersensitivity to boron or mannitol, or compounds containing these components
19. Vaccinated with live, attenuated vaccines within 4 weeks of the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jatin J. Shah, MD, Principal Investigator — UT MD Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: May 10, 2012 to February 08, 2013. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the fourteen participant enrolled, three were screen failures and not enrolled on the study.
Groups:
- Siltuximab + Bortezomib + Lenalidomide: Induction of Lenalidomide 25 mg orally Days 1-14; Bortezomib 1.3 mg/m^2 intravenous Days 1, 4, 8 and 11; Dexamethasone 20 mg orally Days 1, 2, 4, 5, 8, 9, 11, 12. Siltuximab 11 mg/kg intravenous Day 1. If delayed transplant, induction therapy continued up to 2 cycles beyond achieving a CR/nCR then transition to maintenance therapy (Lenalidomide at last tolerated dose Day 1-21 every 28 days for up to 12 months and then may be reduced to 10 mg). Siltuximab 11 mg/kg intravenous every 21 days, or maximum tolerated dose from induction therapy. Bortezomib at last tolerated dose Day 1 and Day 8 Dexamethasone at last tolerated dose or 20 mg weekly.
Period: Overall Study
Arm/Group | Siltuximab + Bortezomib + Lenalidomide
Started | 11
Completed | 8
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Siltuximab + Bortezomib + Lenalidomide
Number analyzed (Participants) | 11
Age, Continuous [Median (Full Range); unit: years] | 62 [47 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Siltuximab
Description: Maximum tolerated dose (MTD) defined as follows: At first dose level, if greater than 1 out of 3 patients or greater than 1 out of 6 patients experience dose limiting toxicity (DLT), the dose level exceeds the maximum tolerated dose (MTD). Dose limiting toxicity (DLT) defined as toxicities graded in severity according to the guidelines outlined in the NCI-Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0.
Time Frame: 21 days
Measure: Number; unit: mg/kg
Arm/Group | Siltuximab + Bortezomib + Lenalidomide
Number analyzed (Participants) | 6
mg/kg | 8.3

2. Secondary Outcome: Number of Participants With Response
Description: Overall response defined as number of participants with International Myeloma Working Group Uniform Response Criteria: Complete Response (CR): Negative immunofixation serum & urine, Disappearance soft tissue plasmacytomas & =/<5% plasma cells in bone marrow; Stringent Complete Remission: CR + Normal Normal free light chain (FLC) ratio & Absence clonal cells in bone marrow by Immunohistochemistry/ immunofluorescence; Very Good Partial Response (VGPR): Serum & urine M-protein detectable by immunofixation but not on electrophoresis or 90%> reduction in serum M-protein +urine M-protein level <100mg per 24 hour; Partial Remission (PR): =/>50% reduction serum M-protein & reduction in 24-hour urinaryMprotein by >90% or to < 200mg per 24 hour, =/>50% reduction of serum M-protein & reduction in 24-hour urinary Mprotein by >90%/or <200mg, and if present at baseline, a >50% reduction in size of soft tissue plasmacytomas; Stable Disease: Not CR, VGPR, PR Or Progressive disease
Time Frame: Evaluated after eight cycles of 21 days.
Measure: Number; unit: participants
Arm/Group | Siltuximab + Bortezomib + Lenalidomide
Number analyzed (Participants) | 11
participants
  Complete Remission (CR) | 2
  Stringent Complete Remission | 0
  Very good partial remission (VGPR) | 2
  Partial Remission (PR) | 6
  Stable Disease | 0

ADVERSE EVENTS:
Time Frame: Adverse event collection during the first cycle of 28-day study drug administration. Overall collection period: May 2012 to February 2013.
Arm/Group | Siltuximab + Bortezomib + Lenalidomide
Serious Adverse Events (participants affected / at risk) | 3/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab + Bortezomib + Lenalidomide (N=11)
Hematuria (Renal and urinary disorders) | 1
Lung infection (Infections and infestations) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Siltuximab + Bortezomib + Lenalidomide (N=11)
Anemia (Blood and lymphatic system disorders) | 11
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 11
Lymphopenia (Blood and lymphatic system disorders) | 10
Leukopenia (Blood and lymphatic system disorders) | 11
Leukocytosis (Blood and lymphatic system disorders) | 1
Alanine Aminotransferase Increased (ALT) (Metabolism and nutrition disorders) | 6
Alanine Aminotransferase Decreased (ALT) (Metabolism and nutrition disorders) | 1
Aspartate Aminotransferase Increased (AST) (Metabolism and nutrition disorders) | 4
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 4
Alkaline Phosphatase, Decreased (Metabolism and nutrition disorders) | 2
Blood Bilirubin Increased (Metabolism and nutrition disorders) | 5
Blood urea nitrogen (BUN), Decreased (Metabolism and nutrition disorders) | 4
BUN, Increased (Metabolism and nutrition disorders) | 5
Chloride, Decreased (Metabolism and nutrition disorders) | 2
Chloride, Increased (Metabolism and nutrition disorders) | 5
Creatinine, Increased (Metabolism and nutrition disorders) | 6
Creatinine, Decreased (Metabolism and nutrition disorders) | 5
Hyperalbuminemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 3
Hyperpophosphatemia (Metabolism and nutrition disorders) | 6
Hyperuricemia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypoglycemia (Metabolism and nutrition disorders) | 5
Hypophosphatamia (Metabolism and nutrition disorders) | 4
Hypouricemia (Metabolism and nutrition disorders) | 5
Hypocalcemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 4
Lactate dehydrogenase (LDH), Decreased (Metabolism and nutrition disorders) | 2
LDH, Increased (Metabolism and nutrition disorders) | 7
Protein, Decreased (Metabolism and nutrition disorders) | 6
Protein, Increased (Metabolism and nutrition disorders) | 5
TSH, Increased (Metabolism and nutrition disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Allergic Reaction (Immune system disorders) | 1
Anxiety (Nervous system disorders) | 1
Bone Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 1
Blurred Vision (Eye disorders) | 7
Chest Pain (General disorders) | 1
Constipation (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Cramps (Calf) (Musculoskeletal and connective tissue disorders) | 1
Dehydration (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 6
Dysgeusia (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 8
Dry Eye (Eye disorders) | 8
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 1
Edema: Limbs (General disorders) | 10
Edema: Trunk (General disorders) | 1
Eye Redness (Eye disorders) | 1
Eye Irritation (Eye disorders) | 1
Fatigue (General disorders) | 11
Facial Drooping (left) (Musculoskeletal and connective tissue disorders) | 1
Fever (Investigations) | 1
Flatulence (Gastrointestinal disorders) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hot Flashes (Endocrine disorders) | 1
Infections and Infestations: Head Boils (Infections and infestations) | 1
Insomnia (General disorders) | 1
Memory Impairment (Nervous system disorders) | 4
Mood Changes (Nervous system disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Muscular & connective tissue Disorder- Other: Muscle Pain (Musculoskeletal and connective tissue disorders) | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Pain (Generalized) (General disorders) | 3
Pain in Extremity (General disorders) | 4
Palpitations (Cardiac disorders) | 1
Paresthesia (Nervous system disorders) | 8
Peripheral Sensory Neuropathy (Nervous system disorders) | 3
Pneumonia (Infections and infestations) | 1
Post Nasal Drip (Immune system disorders) | 2
Progressive Neuropathy (Nervous system disorders) | 1
Rash (Maculo- Papular) (Skin and subcutaneous tissue disorders) | 4
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Soreness (Bilateral) (General disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Upper Respiratory Infection (Infections and infestations) | 3
Urinary Incontinence (Renal and urinary disorders) | 1
Testicular pain (Reproductive system and breast disorders) | 1
Thromboembolic event (Vascular disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 2
Vomiting (Gastrointestinal disorders) | 3
Watering Eyes (Eye disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes